CLINICAL TRIAL: NCT06652932
Title: Acute Effects of Low Temperature Exposure on Respiratory Health in Healthy Young Adults: A Randomized Controlled Study
Brief Title: Acute Effects of Low Temperature Exposure on Respiratory System
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Renjie Chen, Professor, Fudan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: IRB#2024-10-1166
Record Dates: First submitted 2024-10-15; First posted 2024-10-22 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Lung Function
Keywords: Low temperature; Randomized controlled trial; Lung function
MeSH Terms: interventions — Cold Temperature; Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low temperature (15℃) group (Experimental): Subjects in the exposure group will be exposed to low temperature (15℃) for about 2 hours in a chamber.
  Interventions: Other: Low temperature (15°C) group
- Moderate temperature (22℃) group (Experimental): Subjects in the exposure group will be exposed to moderate temperature (22℃) for about 2 hours in a chamber.
  Interventions: Other: Moderate temperature (22°C) group

INTERVENTIONS:
Other: Low temperature (15°C) group — The exposure group will be exposed to low temperature (15°C) in a chamber for about 2 hours, resting during the whole periods.
  Arms: Low temperature (15℃) group
Other: Moderate temperature (22°C) group — The exposure group will be exposed to thermoneutral temperature (22°C) in a chamber for about 2 hours, resting during the whole periods.
  Arms: Moderate temperature (22℃) group

SUMMARY:
This is a randomized controlled human exposure crossover study. Investigators aims to assess the acute effects of low-temperature exposure on respiratory health and the underlying mechanisms.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled human exposure crossover study among about 40 healthy young adults in Shanghai, China. Each subject will be exposed twice: once to the low temperature (15℃) and once to the moderate temperature (22℃) in a chamber for about 2 hours. During the exposure session, each subject will be requested to rest. Health examinations will be conducted immediately prior to exposure, during the period of exposure, and after exposure. Health examinations include lung function tests and exhaled breath test. Investigators plan to collect blood, pharyngeal secretion, exhaled breath condensate and urine samples.

ELIGIBILITY:
Inclusion Criteria:

* Living in Shanghai during the study period;
* Body mass index > 18.5 and ≤ 28;
* right-handed;
* receiving or having received higher education;
* with the ability to read and understand Chinese smoothly.

Exclusion Criteria:

* Smoking and alcohol abuse;
* Current drug and dietary supplements intake;
* Subjects with allergic diseases, such as allergic rhinitis, allergic asthma, and atopy;
* Subjects with cardiovascular diseases, such as congenital heart disease, pulmonary heart disease, and hypertension;
* Subjects with respiratory diseases, such as asthma, chronic bronchitis, and chronic obstructive pulmonary disease;
* Subjects with chronic diseases, such as diabetes, chronic hepatitis, and kidney disease;
* Subjects who have a history of major surgery due to the cardiovascular, cerebrovascular, respiratory, or neurological diseases;
* Subjects with neurologic disorders, such as stroke, traumatic brain injury, epilepsy, and schizophrenia;
* Abnormal spirometry (FEV1 and FVC ≤ 75% of predicted and FEV1/FVC ≤ 0.65);
* Subjects with color vision disabilities.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2024-11-16 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of forced expiratory volume in the first second (FEV1) | The tests will be conducted at 12:30 A.M. (half an hour before exposure) and 3:30 P.M. (half an hour after the exposure)
  Investigators plan to measure the changes of the forced expiratory volume in 1 s (FEV1) using a smart spirometer (Model A1, BreathHome, China) supervised by professional medical staff. Before the pulmonary function test, subjects will practice several times by themselves. During the examination, each subject stands and clamps the nose clip, and repeats the test, with the best result as the criterion. FEV1 reflect pulmonary function.
Changes of forced vital capacity (FVC) | FVC will be examined at 12:30 A.M. (half an hour before exposure) and 3:30 P.M. (half an hour after the exposure)
  Investigators plan to measure the changes of forced vital capacity (FVC) using a portable spirometer (Jaeger Master screen V5.01; CareFusion). FVC reflects the expiratory resistance of large airways.
Changes of peak expiratory flow rate (PEF) | FVC will be examined at 12:30 A.M. (half an hour before exposure) and 3:30 P.M. (half an hour after the exposure)
  Investigators plan to measure the changes of peak expiratory flow (PEF) using a portable spirometer (Jaeger Master screen V5.01; CareFusion). PEF reflects airway patency and respiratory muscle strength.
Changes of maximum expiratory flow rate at 25% vital capacity (MEF25) | MEF25 will be examined at 12:30 A.M. (half an hour before exposure) and 3:30 P.M. (half an hour after the exposure)
  Investigators plan to measure the changes of maximum expiratory flow rate at 25% vital capacity. MEF25% reflects the early stage of expiratory flow rate.
Changes of maximum expiratory flow rate at 50% vital capacity (MEF50) | MEF50 will be examined at 12:30 A.M. (half an hour before exposure) and 3:30 P.M. (half an hour after the exposure)
  Investigators plan to measure the changes of maximum expiratory flow rate at 50% vital capacity using a portable spirometer (Jaeger Master screen V5.01; CareFusion). MEF50 reflects the interim stage of expiratory flow rate.
Changes of maximum expiratory flow rate at 75% vital capacity (MEF75) | MEF75 will be examined at 12:30 A.M. (half an hour before exposure) and 3:30 P.M. (half an hour after exposure)
  Investigators plan to measure the changes of maximum expiratory flow rate at 50% vital capacity (MEF75%) using a portable spirometer (Jaeger Master screen V5.01; CareFusion). MEF75 reflects the terminal stage of expiratory flow rate.

SECONDARY OUTCOMES:
Changes of fractional exhaled nitric oxide (FeNO) | FeNO will be examined half an hour before exposure and half an hour after exposure
  Investigators plan to measure the changes of fractional exhaled nitric oxide using FeNO monitor (NIOX; Aerocrine AB, Solna, Sweden). FeNO reflects airway inflammation level
Changes of fractional concentration of carbon monoxide (FeCO) | FeCO will be examined at 12:30 A.M. (half an hour before exposure) and 3:30 P.M. (half an hour after the exposure)
  Investigators plan to measure the changes of fractional concentration of carbon monoxide using Pico Smokerlyzer. FeCO reflects level of carboxyhemoglobin in blood.
Changes of skin temperature | Wrist skin temperature will be measured at 1:00 P.M. to 3:00 P.M. on the day of the exposure session
  The changes of wrist skin temperature will be measured

OTHER OUTCOMES:
Differences in protein levels detected in blood Clara cell protein (CC16) between the two exposures | CC16 will be examined at 1:00 P.M. and 4:00 P.M. (one hour after the exposure) on the day of the exposure session
  Investigators plan to measure the changes of Clara cell protein using enzyme linked immunosorbent assay (ELISA). Clara cell protein (CC16) indicate lung epithelial injury.
Differences in protein levels detected in blood chitinase-3-like protein 1 (YKL-40) between the two exposures | YKL-40 will be examined at 1:00 P.M. and 4:00 P.M. (one hour after exposure) on the day of the exposure session
  Investigators plan to measure the changes of chitinase-3-like protein 1 protein using enzyme linked immunosorbent assay (ELISA). YKL-40 represents airway inflammation and remodeling.
Differences in protein levels detected in blood Surfactant Protein-D (SP-D) between the two exposures | SP-D will be examined at 1:00 P.M. and 4:00 P.M. (one hour after exposure) on the day of the exposure session
  Investigators plan to measure the changes of Surfactant Protein-D protein using enzyme linked immunosorbent assay (ELISA). SP-D represents pulmonary injury.
Differences in respiratory microbiota detected in pharyngeal secretion between the two exposures | Respiratory microbiota will be detected at 3:30 A.M. (half an hour after exposure) on the day of the exposure session
  differential respiratory microbiota in pharyngeal secretion related to low temperature exposure will be detected by integrating microbial 16S rRNA sequencing and non-targeted metabolomics.
Differences in metabolic profiling detected in exhaled breath condensate between the two exposures | Metabolic profiling in exhaled breath condensate will be detected at 4:00 P.M. (1 hour after the exposure session)
  The differential metabolic profiling in exhaled breath condensate related to low temperature exposure will be detected by mass spectrometry-based non-targeted metabolomics.

CONTACTS AND LOCATIONS:
Overall Officials: Haidong Kan, PhD, Study Director — Fudan University
Locations (1):
- Department of Environmental Health, School of Public Health, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-10-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT06652932/SAP_000.pdf